CLINICAL TRIAL: NCT02667119
Title: Treating Co-Occurring PTSD and Substance Abuse in High-Risk Transition Age Youth
Brief Title: Integrated Treatment for Posttraumatic Stress Disorder and Substance Abuse in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kristyn Zajac, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-101-2; K23DA034879 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Substance Use Disorder; Posttraumatic Stress Disorder
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure + Contingency Management (Experimental): Standard services plus Prolonged Exposure and Contingency Management
  Interventions: Behavioral: Prolonged Exposure with Contingency Management; Behavioral: Standard Care
- Standard Care (Active Comparator): Standard substance abuse treatment services
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Prolonged Exposure with Contingency Management — Prolonged Exposure therapy for posttraumatic stress disorder includes psychoeducation, breathing retraining, in vivo exposure, and imaginal exposure.
  Contingency Management for substance abuse disorders: participants will have the chance to win prizes for each negative urine drug screen/breathalyzer provided.
  Arms: Prolonged Exposure + Contingency Management
Behavioral: Standard Care — Standard care will consist of treatment as usual in a community-based substance use treatment center.

SUMMARY:
The purpose of the study is to determine the safety and efficacy of an integrated treatment for substance abuse and posttraumatic stress disorder for young adults. The integrated treatment includes two established psychosocial treatments for substance abuse (Contingency Management) and posttraumatic stress disorder (Prolonged Exposure therapy).

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old
* meets diagnostic criteria for substance use disorder
* meets diagnostic criteria for full or subthreshold posttraumatic stress disorder
* currently able to provide a urine drug screen that is negative for cocaine, prescription opiates, and non-prescribed methadone or provided this type of screen in the past 60 days
* speaks English

Exclusion Criteria:

* significant cognitive impairment or serious uncontrolled psychiatric problem (other than posttraumatic stress disorder)
* in recovery from pathological gambling or current pathological gambling diagnosis
* in a current domestic violence relationship

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04; Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristyn Zajac, PhD, Principal Investigator — UConn Health
Locations (3):
- United States (3):
  - UConn Health, Farmington, Connecticut
  - The Village for Families and Children - Adult Services, Hartford, Connecticut
  - Farrell Treatment Center, New Britain, Connecticut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zajac K, Sheidow AJ, Davis M. Juvenile Justice, Mental Health, and the Transition to Adulthood: A Review of Service System Involvement and Unmet Needs in the U.S. Child Youth Serv Rev. 2015 Sep 1;56:139-148. doi: 10.1016/j.childyouth.2015.07.014. PMID 26273119
- [Background] Zajac K, Randall J, Swenson CC. Multisystemic Therapy for Externalizing Youth. Child Adolesc Psychiatr Clin N Am. 2015 Jul;24(3):601-16. doi: 10.1016/j.chc.2015.02.007. Epub 2015 Mar 29. PMID 26092742

RESULTS

PARTICIPANT FLOW:
Groups:
- Prolonged Exposure + Contingency Management: Standard services plus Prolonged Exposure and Contingency Management
  Prolonged Exposure with Contingency Management: Prolonged Exposure therapy for posttraumatic stress disorder includes psychoeducation, breathing retraining, in vivo exposure, and imaginal exposure.
  Contingency Management for substance abuse disorders: participants will have the chance to win prizes for each negative urine drug screen/breathalyzer provided.
  Standard Care: Standard care will consist of treatment as usual in a community-based substance use treatment center.
Period: Overall Study
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Started | 14 | 13
Completed | 11 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.93 (1.89) | 22.46 (2.11) | 22.70 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 13 | 6 | 19
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
National Stressful Events PTSD Scale [Mean (Standard Deviation); unit: scores on a scale] — Presented as an item mean. Minimum score = 1. Maximum score = 5. Higher equals worse symptoms.
  scores on a scale | 3.26 (.58) | 2.82 (.58) | 3.05 (.70)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Posttraumatic Stress Disorder Symptoms as Measured by the National Stressful Events PTSD Scale
Description: National Stressful Events Posttraumatic Stress Disorder Short Scale. Outcome is presented as a mean item score. Minimum value = 1, Maximum value = 5. Higher scores mean worse outcomes (more severe symptoms).
Time Frame: Baseline and 3-months post-baseline
Population: Two participants from the Prolonged Exposure + Contingency Management group and one participant from the Standard Care group did not complete assessments at 3 months post-baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 12 | 12
score on a scale | 1.92 (.92) | 2.61 (1.15)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Compared the two groups at 3 months post-baseline; Test type: Superiority; p = .041, ANCOVA; Controlled for baseline scores on the National Stressful Events PTSD Scale; F = 4.75

2. Primary Outcome: Change in Severity of Posttraumatic Stress Disorder Symptoms as Measured by the National Stressful Events PTSD Scale
Description: as for outcome 1
Time Frame: Baseline and 6-month post-baseline
Population: Three participants from the Prolonged Exposure + Contingency Management group did not complete assessments at 6 months post-baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 11 | 13
score on a scale | 1.64 (.65) | 2.29 (.93)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Test type: Superiority; p = .016, ANCOVA; Controlled for baseline score on the National Stressful Events PTSD Scale; F = 6.89

3. Primary Outcome: Longest Duration of Abstinence From Illicit Drugs (Physiological Measure - Urine Drug Screens)
Description: Illicit drug use is assessed twice weekly during the 10 week treatment period. Longest duration of abstinence is calculated as the longest time period in weeks of consecutive negative urine drug screens for illicit drugs during the 10 weeks of treatment.
Time Frame: 10 week treatment period
Population: Full sample was included
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 14 | 13
weeks | 4.29 (3.73) | 1.77 (2.05)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Test type: Superiority; p = .04, t-test, 2 sided; t = -2.19

4. Secondary Outcome: Change in Severity of Depression Symptoms as Measured by the Center for Epidemiological Studies-Depressed Mood Scale
Description: Center for Epidemiological Studies-Depressed Mood. Minimum value = 0. Maximum value = 60. Higher scores mean worse outcomes (more severe symptoms).
Time Frame: Baseline and 3-month post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 12 | 12
score on a scale | 17.75 (13.75) | 23.33 (17.92)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Test type: Superiority; p = .148, ANCOVA — Controlling for baseline score on the Center for Epidemiological Studies-Depressed Mood scale; F = 2.25

5. Secondary Outcome: Change in Severity of Depression Symptoms as Measured by the Center for Epidemiological Studies-Depressed Mood Scale
Description: as for outcome 4
Time Frame: Baseline and 6-month post-baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 11 | 13
score on a scale | 14.64 (10.70) | 21.69 (15.14)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Test type: Superiority; p = .043, ANCOVA; Controlling for baseline score on the Center for Epidemiological Studies-Depressed Mood scale; F = 4.64

6. Secondary Outcome: Change in Quality of Life as Measured by the Quality of Life Scale
Description: Quality of Life Scale. Minimum value = -6. Maximum value = +6. Score is an item mean. Higher scores mean better outcomes.
Time Frame: Baseline and 3-month post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 12 | 12
score on a scale | 1.66 (1.94) | 1.36 (2.01)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Test type: Superiority; p = .250, ANCOVA — Controlling for baseline score on the Quality of Life Scale; F = 1.40

7. Secondary Outcome: Change in Quality of Life as Measured by the Quality of Life Scale
Description: as for outcome 6
Time Frame: Baseline and 6-month post-baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
Number analyzed (Participants) | 11 | 13
score on a scale | 1.44 (1.54) | 1.33 (1.64)
Statistical Analysis 1: Comparison: Prolonged Exposure + Contingency Management vs Standard Care; Test type: Superiority; p = .508, ANCOVA; Controlling for baseline score on the Quality of Life Scale; F = .45

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Prolonged Exposure + Contingency Management | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/14 | 4/13
Other Adverse Events (participants affected / at risk) | 4/14 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure + Contingency Management (N=14) | Standard Care (N=13)
Inpatient substance use treatment (General disorders) | 1 (1) | 3 (3)
Suicidal ideation (life threatening) (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure + Contingency Management (N=14) | Standard Care (N=13)
Suicidal ideation (not life threatening) (Psychiatric disorders) | 3 (3) | 3 (4)
Emergency room visit (General disorders) | 2 (2) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT02667119/Prot_SAP_000.pdf